CLINICAL TRIAL: NCT00137176
Title: EARLY IFNb-1a (Rebif) and Atorvastatin (Lipitor) Combination Therapy of Isolated Clinical Syndrome Suggestive of Multiple Sclerosis
Brief Title: EARLY IFNb-1a and Atorvastatin Combination Therapy of Isolated Clinical Syndrome Suggestive of Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Silva Markovic-Plese, UNC Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 04-NEUR-293
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2009-06-23 (Estimated); Status verified 2009-06

CONDITIONS: Multiple Sclerosis
Keywords: Clinically Isolated Syndrome
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rebif + Lipitor (Experimental)
  Interventions: Drug: Rebif

INTERVENTIONS:
Drug: Rebif — Rebif 44mcg TIW

SUMMARY:
The primary purpose is to determine the changes in gene expression induced by IFNb-1a (Rebif) and atorvastatin (Lipitor) combination therapy in patients with an isolated clinical syndrome suggestive of multiple sclerosis (MS), to identify markers of therapeutic response, and to predict patients' clinical response based on their in vitro response to this combination therapy measured by the gene expression levels in activated peripheral blood mononuclear cells (PBMCs).

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic neurologic disease, characterized pathologically by focal areas of inflammation, demyelination, axonal injury and degeneration in the central nervous system. MS follows several different disease courses. Approximately, 90% of patients have a relapsing form of the disease. We propose that atorvastatin (Lipitor) may enhance the immunomodulatory effects of INFb-1a (Rebif) in patients with clinically isolated neurological syndrome suggestive of MS. This combination may be more effective in preventing development of definitive relapsing-remitting MS if administered early in the course of the disease. The study will identify markers of disease activity that are selectively affected by this combination therapy. Identified markers may be used in future clinical trials to predict patient's clinical response and to monitor the response to treatment as a secondary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with isolated clinical syndrome suggestive of MS
* At least three out of four magnetic resonance imaging (MRI) findings on the initial scan:

  * One Gd-enhancing lesion or nine T2 hyperintense lesions;
  * At least one infratentorial lesion;
  * At least one juxtacortical lesion; and
  * At least three periventricular lesions.
* Expanded Disability Status Scale (EDSS) 0-5.5
* 18 to 60 years of age
* At least one relapse in previous 12 months

Exclusion Criteria:

* Patients with a diagnosis of clinically definitive relapsing-remitting (RR) MS, secondary progressive, or primary progressive MS.
* Patients who have ever been treated with mitoxantrone, cytoxan, cyclophosphamide, or total lymphoid irradiation (TLI).
* Patients treated with IFNb-1a, IFNb-1b, glatiramer acetate, intravenous immunoglobulins (IVIg), plasma exchange, methotrexate, or azathioprine in the previous 3 months.
* Patients treated with intravenous or oral steroids within 30 days prior to baseline MRI.
* Patients who have been treated with statins in the previous 3 months.
* Pregnant or breast-feeding women.
* Patients with a history of severe cardiac, hepatic, pulmonary, gastrointestinal, or renal disease.
* Abnormal baseline blood tests including alanine transaminase (ALT) or aspartate transaminase (AST) greater than twice the upper limit of normal

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-10; Primary Completion 2007-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To determine the effects of IFNb-1a plus atorvastatin versus IFNb-1a plus placebo on the gene expression in peripheral blood mononuclear cells (PBMCs) derived from patients with isolated clinical syndrome suggestive of MS | 2 years
To identify markers of therapeutic response and to predict patients' clinical response based on their in vitro response to this combination therapy measured by the gene expression levels in activated PBMCs | 2 years

SECONDARY OUTCOMES:
evaluate safety and efficacy of combination therapy with Rebif and Lipitor in patients with clinicayy isolated syndrome suggestive of MS. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Silva Markovic-Plese, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina-Chapel Hill MS Clinic Within the Neuroscience Hospital, Chapel Hill, North Carolina, United States